CLINICAL TRIAL: NCT05562934
Title: A Multi-center, Randomized, Double-blind, Parallel-group, 20-week Dose-finding Study to Evaluate Efficacy, Safety, and Tolerability of XXB750 in Patients With Resistant Hypertension
Brief Title: An Efficacy, Safety, Tolerability and Dose Finding Study of XXB750 in Resistant Hypertension Patients.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CXXB750B12201; 2021-005738-41 (EudraCT Number)
Record Dates: First submitted 2022-09-28; First posted 2022-10-03 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Resistant Hypertension
Keywords: hypertension; resistant hypertension; rHTN; not controlled hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: The planned duration of treatment is 12 weeks per participant. Participants may be discontinued from treatment earlier due to unacceptable adverse events, disease progression and/or if treatment is discontinued at the discretion of the investigator or the participant. Following the conclusion of the 12-week Randomized Treatment Period, participants will enter an 8-week Safety Follow-up Period in which participants may be treated at the discretion of the investigator taking into account that their blood pressure may still be affected by the study treatment for some time after its discontinuation, especially those who were randomized to XXB750.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants, investigator staff, persons performing the assessments and blinded clinical research associate (CRA) monitoring study conduct remained blinded to the identity of the treatment from the time of randomization until database lock. The study site pharmacist/nurse or other designated qualified site personnel who prepares the study drug and the unblinded clinical research associates (CRA monitoring drug supply and preparation) remained unblinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose 1 (Experimental): Lowest dose
  Interventions: Biological: XXB750 drug
- Dose 2 (Experimental): Dose 2
  Interventions: Biological: XXB750 drug
- Dose 3 (Experimental): Dose 3
  Interventions: Biological: XXB750 drug
- Dose 4 (Experimental): Highest dose
  Interventions: Biological: XXB750 drug
- Dose 5 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: XXB750 drug — SC injection
  Arms: Dose 1; Dose 2; Dose 3; Dose 4
Other: Placebo — SC injection
  Arms: Dose 5

SUMMARY:
The purpose of this 20-week randomized double-blind study in patients with resistant hypertension (rHTN) is to evaluate the efficacy, safety, and tolerability, of different doses of XXB750 administered as subcutaneous (SC) injections, compared to placebo. Since all study participants will be patients with rHTN, all study treatments will be given on top of maximally tolerated background antihypertensive therapy recommended by international guidelines for treatment of HTN (i.e., a thiazide or a thiazide-like diuretic, an angiotensin converting enzyme inhibitor (ACEi) or an angiotensin receptor blocker (ARB), and a long-acting dihydropyridine calcium channel blocker (CCB).

DETAILED DESCRIPTION:
Subjects will enter run-in period which lasts for approximately 2 weeks. The study duration is for 20 weeks during which each participant will receive a total of 3 doses of study medication (in addition to 1 dose of study medication during run-in). Participants will be followed to monitor their safety for an additional 8 weeks during which time no active study medication will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants who are ≥ 18 years old.
2. Signed informed consent prior to participation in the study.
3. Apparent rHTN at screening (Visit 1) defined as uncontrolled BP with an office msSBP ≥ 140 mmHg despite treatment with stable (i.e., unchanged for ≥4 weeks), optimal or maximally tolerated doses of three or four antihypertensive drugs of different classes, including an ACEI/ARB, a long-acting dihydropyridine CCB, and a thiazide or thiazide-like diuretic. Participant with documented intolerance to any doses of CCBs may be eligible if receiving another class of antihypertensive medication at an optimal or maximally tolerated dose (referred to as triple background antihypertensive therapy. An optimal dose is defined as the highest dose taking in to account participant's documented comorbidities and tolerability per investigator's clinical judgment.
4. Mean 24hr SBP ≥135 mmHg (measured by ABPM) at the end-of Run-in-Visit (Visit 30) on treatment with optimal or maximally tolerated doses of an ACEI/ARB, a long-acting dihydropyridine CCB (or a suitable alternative in case of intolerance per inclusion criterion above), and a thiazide or thiazide-like diuretic.

Exclusion Criteria:

1. Subjects with the following blood pressures at the specified time points are not eligible to participate in the study:

   1. Office msSBP <140 mmHg at Visit 20 OR
   2. Office msSBP ≥180 mmHg or office msDBP ≥110 mmHg at the end-of-run-in visit (Visit 30) OR
   3. 24h mean SBP >170 mmHg or 24h mean DBP >105mmHg measured by ABPM at the end of the run-in (Visit 30).
2. Known history of secondary hypertension (moderate-to-severe obstructive sleep apnea without receiving CPAP therapy (either face mask or nasal device), renovascular hypertension, primary aldosteronism, pheochromocytoma, Cushing syndrome, aortic coarctation or other cause of secondary hypertension).
3. Estimated GFR <30 mL/min/1.73m2 using CKD-Epi equation at screening (Visit 1) or at end-of-run-in visit (Visit 30).
4. Serum potassium >5.0 mmol/L (or equivalent plasma potassium value) at screening or end-of-run-in visit (Visit 30).
5. Current therapy with a mineralocorticoid receptor antagonist (MRA) or sacubitril/valsartan or received an MRA or sacubitril/valsartan within the 4 weeks prior to screening.
6. Type I diabetes mellitus or uncontrolled Type II diabetes (defined as a plasma HbA1c ≥9%)
7. Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), high-grade AV block (e.g., Mobitz type II and third-degree AV block in absence of a pacemaker) within 6 months of screening according to investigator's judgement.
8. Chronic non-paroxysmal atrial fibrillation.
9. Acute myocardial infarction (AMI) or unstable angina, or any history of ischemic or hemorrhagic stroke within 12 months of screening; or any percutaneous coronary intervention (PCI) or coronary artery bypass graft (CABG) within 12 months of screening
10. History of a renal denervation procedure.
11. Mid-arm circumference ≥44 cm. The cuff should snugly fit on the arm with out the margins of cuff overhanging arm musculature.
12. Patients with history of hospitalisation for hypertensive emergencies characterised by severe hypertension (usually grade 3) associated with funduscopic changes (flame haemorrhages and/or papilloedema), microangiopathy, disseminated intravascular coagulation, encephalopathy, acute aortic dissection, acute myocardial ischaemia, or acute heart failure any time prior to screening or hospitalisation for non-emergent/non-urgent uncontrolled hypertension without target organ damage within 3 months prior to screening
13. Receiving more than 4 antihypertensive medications.
14. Night shift workers.
15. History of presence of any other disease where the life expectancy is less than 3 years.
16. History of malignancy of any organ system (other than localized basal or squamous cell carcinoma of the skin or localized prostate cancer), treated or untreated, within the past 3 years, regardless of whether there is evidence of local recurrence or metastases.
17. Evidence of hepatic disease as determined by any one of the following: SGOT (AST) or SGPT (ALT) values exceeding 3x the upper limit of normal (ULN), or bilirubin >1.5 mg/dl at Visit 1.
18. Use of other investigational drugs at the time of enrollment, or within 30 days or 5 half-lives of enrollment, whichever is longer.
19. History of drug abuse or alcohol dependency.
20. Lacking the ability to comprehend or follow instructions, or for any reason in the opinion of the investigator, a participant that would be unlikely or unable to comply with study protocol.
21. Concurrent enrollment in any other investigational drug or device trial (participation in non-interventional registries is acceptable).
22. Requiring prolonged/regular use of NSAIDs except for prophylactic use of low dose aspirin up to 325 mg QD or other prohibited medications during of the study (i.e., required use for longer than 1 week).
23. Pregnant, nursing or planning to become pregnant (documented negative pregnancy test required within a maximum of 7 days prior to enrollment of all women of childbearing potential). Documentation of highly effective contraception is also required for women of childbearing potential (see below).

    Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception while taking study treatment and for 3 months after stopping medication. Highly effective contraception methods include:
    * Total abstinence (when this is in line with the preferred and usual lifestyle of the participant. Periodic abstinence (e.g. calendar, ovulation, symptom-thermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or bilateral tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment.
    * Male sterilization (at least 6 months prior to screening). For female participants on the study, the vasectomized male partner should be the sole partner for that participant.
    * Use of oral, (estrogen and progesterone), injected, or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate < 1%), for example hormone vaginal ring or transdermal hormone contraception.

    In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age-appropriate history of vasomotor symptoms). Women are considered not of childbearing potential if they are post-menopausal or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy or bilateral tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential.

    If local regulations deviate from the contraception methods listed above to prevent pregnancy, local regulations apply and will be described in the ICF.
24. History of hypersensitivity to any of the study drugs, excipients or drugs of similar class.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2024-07-02 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (72):
- United States (18):
  - Pinnacle Research Group Llc, Anniston, Alabama
  - Parkway Medical Center, Birmingham, Alabama
  - Clinical Trials Research Sacramento, Sacramento, California
  - Orange County Research Center, Tustin, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Canvas Clinical Research, Lake Worth, Florida
  - Inpatient Research Clinical LLC, Miami Lakes, Florida
  - Cardiology Partners Clinical Research Institute, Wellington, Florida
  - American Clinical Trials, Acworth, Georgia
  - Alliance for Multispecialty Resrch, Wichita, Kansas
  - Anderson Medical Research, Ft. Washington, Maryland
  - Capitol Cardiology Associates, Lanham, Maryland
  - MD Medical Research, Oxon Hill, Maryland
  - NexGen Research, Lima, Ohio
  - The Research Center of the Upstate, Greenville, South Carolina
  - Tennessee Center For Clinical Trials, Tullahoma, Tennessee
  - Manassas Clinical Research Center, Manassas, Virginia
  - Dominion Medical Associates, Richmond, Virginia
- Australia (2):
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Perth, Western Australia
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Vienna
- Bulgaria (2):
  - Novartis Investigative Site, Pleven
  - Novartis Investigative Site, Sofia
- China (5):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Baotou, Inner Mongolia
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Qingdao
  - Novartis Investigative Site, Shanghai
- Czechia (2):
  - Novartis Investigative Site, Brandýs nad Labem, Czech Republic
  - Novartis Investigative Site, Prague
- France (4):
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Tours
- Germany (5):
  - Novartis Investigative Site, Elsterwerda, Brandenburg
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Ulm
- Italy (4):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Brescia, BS
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pisa, PI
- Japan (7):
  - Novartis Investigative Site, Chikushino-shi, Fukuka
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Yokosuka, Kanagawa
  - Novartis Investigative Site, Kishiwada, Osaka
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
- Novartis Investigative Site, Amsterdam, North Holland, Netherlands
- Poland (4):
  - Novartis Investigative Site, Gdynia
  - Novartis Investigative Site, Katowice
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Wroclaw
- Slovakia (4):
  - Novartis Investigative Site, Bardejov
  - Novartis Investigative Site, Košice
  - Novartis Investigative Site, Nitra
  - Novartis Investigative Site, Svidník
- Spain (7):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Terrassa, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Valencia
- Taiwan (2):
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (3):
  - Novartis Investigative Site, London, GBR
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Salford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] White WB, Azizi M, Ferdinand K, Cohen DL, Nuhrenberg T, Lefkowitz M, Jiao R, Rizkala AR, Maboudian M, Williams B. Natriuretic Peptide Receptor-1 Agonist for Resistant Hypertension: A Randomized Phase 2 Trial. J Am Coll Cardiol. 2026 Jan 13:S0735-1097(25)10351-3. doi: 10.1016/j.jacc.2025.11.045. Online ahead of print. PMID 41563174
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2799

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 135 investigative sites in 16 countries.
Pre-assignment Details: The study consisted of a screening period of approximately 7 days.
Groups:
- Placebo: Placebo subcutaneous (s.c) every 4 weeks, total of 3 doses.
- XXB750 30 mg: XXB750 30 mg s.c every 4 weeks, total of 3 doses.
- XXB750 60 mg: XXB750 60 mg s.c every 4 weeks, total of 3 doses.
- XXB750 120 mg: XXB750 120 mg s.c every 4 weeks, total of 3 doses.
- XXB750 120 mg/240 mg: XXB750 120 mg s.c at the randomization visit followed by 240 mg s.c at Week 4 and Week 8.
Period: Overall Study
Arm/Group | Placebo | XXB750 30 mg | XXB750 60 mg | XXB750 120 mg | XXB750 120 mg/240 mg
Started | 42 | 32 | 36 | 37 | 42
Completed | 42 | 30 | 35 | 35 | 38
Not Completed | 0 | 2 | 1 | 2 | 4
Not completed — Adverse Event | 0 | 2 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | XXB750 30 mg | XXB750 60 mg | XXB750 120 mg | XXB750 120 mg/240 mg | Total
Number analyzed (Participants) | 42 | 32 | 36 | 37 | 42 | 189
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.14 (10.862) | 58.53 (11.565) | 63.44 (10.191) | 62.41 (11.642) | 60.64 (10.085) | 61.05 (10.863)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 6 | 18 | 13 | 58
  Male | 29 | 24 | 30 | 19 | 29 | 131
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black Or African American | 6 | 7 | 4 | 4 | 6 | 27
  White | 27 | 16 | 24 | 24 | 25 | 116
  Asian | 8 | 5 | 6 | 8 | 10 | 37
  Other | 1 | 4 | 2 | 1 | 1 | 9

OUTCOME MEASURES:

1. Primary Outcome: Dose-response (DR) Relationship of XXB750 With Respect to Change From Baseline in Systolic Blood Pressure (SBP) 24 Hours
Description: To evaluate the efficacy and dose-response relationship of different doses of XXB750 compared to placebo in reducing the mean 24 hours ambulatory systolic blood pressure from baseline at Week 12. Automated arterial BP determinations and pulse rate readings were made with Microlife Watch BP Office 2G, an automated digital BP device. The primary outcome measure was evaluated using an optimally weighted contrast test following the Multiple Comparison Procedure-Modeling (MCP-MOD) methodology. There were five candidate models to capture the shape of the dose-response relationship for XXB750 at Week 12 endpoint. The outcome for the single best candidate model is shown in the Statistical Analysis section.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS): All participants to whom study treatment was assigned by randomization. Only participants with a valid assessment for this endpoint were included.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Placebo | XXB750 30 mg | XXB750 60 mg | XXB750 120 mg | XXB750 120 mg/240 mg
Number analyzed (Participants) | 40 | 25 | 30 | 32 | 36
mmHg | -5.77 [-10.74 to -1.12] | -6.41 [-10.15 to -2.85] | -6.63 [-10.40 to -3.53] | -6.66 [-12.57 to -3.16] | -5.40 [-9.58 to -0.36]
Statistical Analysis 1: Comparison: Placebo vs XXB750 30 mg vs XXB750 60 mg vs XXB750 120 mg vs XXB750 120 mg/240 mg; Test type: Superiority; p = 0.5651, Multiple Comparisons Procedure-MOD — Single best candidate model is the one with the lowest adjusted p-value of the 5 candidate models

2. Secondary Outcome: Change From Baseline in SBP 24 Hours at Week 12 (Difference Between Highest XXB750 Dose and Placebo)
Description: To evaluate the treatment effect of the highest XXB750 dose versus placebo in reducing the mean 24 hours SBP from baseline to Week 12. Automated arterial BP determinations and pulse rate readings were made with Microlife Watch BP Office 2G, an automated digital BP device.
Time Frame: Baseline, Week 12
Population: Full analysis set (FAS): All participants to whom study treatment was assigned by randomization. Only participants from the highest XXB750 dose and placebo with valid measurements are included.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | XXB750 120 mg/240 mg
Number analyzed (Participants) | 40 | 36
mmHg | -6.01 (2.42) | -4.64 (2.49)
Statistical Analysis 1: Comparison: Placebo vs XXB750 120 mg/240 mg; Test type: Superiority; p = 0.6955, ANCOVA; Median Difference (Net) = 1.37, 95% CI 2-sided [-5.48 to 8.21]

3. Secondary Outcome: Change From Baseline in SBP 24 Hours of Average of Week 9 and Week 12 (Difference Between Highest XXB750 Dose and Placebo)
Description: To evaluate the treatment effect of the highest XXB750 dose versus placebo in the dosing interval average of ambulatory SBP as assessed by average of mean 24 hours SBP measured at week 9 and week 12. Automated arterial BP determinations and pulse rate readings were made with Microlife Watch BP Office 2G, an automated digital BP device.
Time Frame: Baseline, Week 9 and Week 12
Population: Full analysis set (FAS): All participants to whom study treatment was assigned by randomization. Only participants from the highest XXB750 dose and placebo with valid measurements (with non-missing observed change from baseline either at Week 9 or Week 12) are included.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Placebo | XXB750 120 mg/240 mg
Number analyzed (Participants) | 40 | 38
mmHg | -5.77 (2.13) | -4.62 (2.21)
Statistical Analysis 1: Comparison: Placebo vs XXB750 120 mg/240 mg; Test type: Superiority; p = 0.7108, ANCOVA; Median Difference (Net) = 1.14, 95% CI 2-sided [-4.90 to 7.18]

4. Secondary Outcome: The Model-based Estimated Percentage of Participants Achieving Blood Pressure (BP) Control
Description: To evaluate the percentage of participants achieving ambulatory BP control defined as mean 24 hours SBP <130 mmHg and mean 24 hours DBP < 80 mmHg with respect to the dose-response relationship of the four XXB750 dose level groups compared to placebo at week 12. Automated arterial BP determinations and pulse rate readings were made with Microlife Watch BP Office 2G, an automated digital BP device. Percentage of participants is derived from dose response analysis, using generalized MCP-Mod methodology for binary data.
Time Frame: Week 12
Population: Full analysis set (FAS): All participants to whom study treatment was assigned by randomization.
Measure: Number; unit: percentage
Arm/Group | Placebo | XXB750 30 mg | XXB750 60 mg | XXB750 120 mg | XXB750 120 mg/240 mg
Number analyzed (Participants) | 40 | 25 | 30 | 32 | 36
percentage | 13.2 | 15.0 | 17.7 | 22.0 | 25.9

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus follow up period, up to a maximum duration of approximately 20 weeks.
Arm/Group | Placebo | XXB750 30 mg | XXB750 60 mg | XXB750 120 mg | XXB750 120 mg/240 mg
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/32 | 0/36 | 0/37 | 0/42
Serious Adverse Events (participants affected / at risk) | 1/42 | 2/32 | 3/36 | 1/37 | 3/42
Other Adverse Events (participants affected / at risk) | 27/42 | 19/32 | 18/36 | 16/37 | 18/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | XXB750 30 mg (N=32) | XXB750 60 mg (N=36) | XXB750 120 mg (N=37) | XXB750 120 mg/240 mg (N=42)
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Osteomyelitis acute (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Exertional rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=42) | XXB750 30 mg (N=32) | XXB750 60 mg (N=36) | XXB750 120 mg (N=37) | XXB750 120 mg/240 mg (N=42)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0
Injection site pain (General disorders) | 0 | 0 | 1 | 0 | 1
Injection site pruritus (General disorders) | 0 | 0 | 0 | 0 | 1
Injection site reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 3 | 2 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0
COVID-19 (Infections and infestations) | 4 | 1 | 0 | 0 | 3
Carbuncle (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infected bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Injection site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Pneumonia aspiration (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 4 | 1 | 0 | 4 | 1
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Burns first degree (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 2 | 0 | 0 | 1
Blood iron abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0
Electrocardiogram PR prolongation (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram ST-T segment elevation (Investigations) | 0 | 0 | 1 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Glucose urine present (Investigations) | 1 | 0 | 1 | 0 | 0
Haematocrit increased (Investigations) | 0 | 1 | 0 | 0 | 0
Haemoglobin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Heart rate abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Heart sounds abnormal (Investigations) | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 1
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 1
Protein urine present (Investigations) | 1 | 0 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 0 | 0 | 1 | 1 | 2
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 3 | 0
Impaired fasting glucose (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Glomus tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 3 | 2 | 1 | 2
Headache (Nervous system disorders) | 1 | 2 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 1 | 0 | 0
Hypotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Vertebral artery occlusion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
Irritability (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Albuminuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Nocturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0 | 1 | 2 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 3 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Skin swelling (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Solar urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 1 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT05562934/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-26): https://cdn.clinicaltrials.gov/large-docs/34/NCT05562934/SAP_001.pdf